CLINICAL TRIAL: NCT03586505
Title: Tolerance to Light for Patients Suffering From Keratitis
Acronym: EBLOUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University of Saint-Etienne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1708072; 2017-A03451-52 (Other: ANSM)
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Keratitis
Keywords: Keratitis; Eye Infection; Photophobia; Red light; Infrared light
MeSH Terms: conditions — Keratitis; Eye Infections; Photophobia

STUDY DESIGN:
Intervention Model Description: Each patient is its own control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light exposure (Experimental): The keratitis eye of the patient is exposed to 6 lights with increasing intensity according to a constant speed.
  The patients switch off the light when the discomfort is too elevated
  Interventions: Device: Light exposure

INTERVENTIONS:
Device: Light exposure — The 6 lights used randomly are :
  * 482nm =standard blue light illumination,
  * 650nm,
  * 675nm,
  * 700nm,
  * 750nm
  * 800nm

SUMMARY:
In order to develop an innovative device to study infectious keratitis, we need to illuminate the cornea of patients suffering from an infectious keratitis with red or near-infrared light. Because of technical reasons the shortest possible wavelength (red) presents advantages.

DETAILED DESCRIPTION:
The aim of this preliminary study is to measure the maximal intensity tolerated during illumination with 6 wavelength corresponding : 2 red, 2 far red and 1 near infrared lights in order to determine the shortest wavelength well tolerated by patients, in comparison with the standard blue light illumination.

ELIGIBILITY:
Inclusion Criteria:

* Social security insurance
* Suspected infectious keratitis (clinically defined. No lab testing required)
* Signed informed consent

Exclusion Criteria:

* Major Blepharospasm
* Aphakia (absence of lens)
* Pregnant woman
* Nursing mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Light intensity | At the inclusion
  For each wavelength, the highest light intensity tolerated by the patient is measured (mWatts/cm² )

SECONDARY OUTCOMES:
Severity of the keratitis | At the inclusion
  It is determined by slit lamp. The result is "severe" or "not severe"

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courrier E, Lambert V, Renault D, Garcin T, Moine B, Herbepin P, Thuret G, Gain P. Tolerance to Light of Patients Suffering From Infectious Keratitis. Cornea. 2021 Jan;40(1):5-11. doi: 10.1097/ICO.0000000000002516. PMID 33038155